CLINICAL TRIAL: NCT06378424
Title: The Effectiveness of Local Dry Cold, Hot and Vibration Applications During Peripheral Intravenous Catheterization Placement in the Emergency Unit
Brief Title: The Effectiveness of Local Dry Cold, Hot and Vibration Applications in Peripheral Intravenous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Associate Professor, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-6/6
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pain Management; Emergency Unit; Diarrhea; Nausea; Vomiting
Keywords: Hot application; cold application; peripheral intravenous catheterization; venous dilation; pain; vibration
MeSH Terms: conditions — Agnosia; Emergencies; Diarrhea; Nausea; Vomiting; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold Application Group (Experimental): Before peripheral intravenous catheterization, dry cold was applied to the application area using a cold gel pack. For this purpose, a 11 x10 cm pack of non-toxic gel was frozen solid in the refrigerator. Because this pack is reusable, it was disinfected before and after each use, and left in the service refrigerator to freeze solid. Attention was paid that it was used in solid form with all individuals.
  Interventions: Other: Cold Application
- Heat Application Group (Experimental): Before peripheral intravenous catheterization, heat of approximately 40-42 o C was applied for 1 minute to the area of the procedure using a hot pack, which is one of the dry heat application methods. The heat application pack has a feature that it can maintain its temperature when taken out of hot water and does not disturb the person when it comes into direct contact with the skin. In order to apply heat to the individuals in this group, a pack of 11 x 19 cm is used. This pack is covered with cloth and contains a non-toxic gel, and is placed in hot water to prepare it for use. Because this pack is reusable, it was disinfected before and after each use.
  Interventions: Other: Heat Application
- Vibration Application Group (Experimental): With individuals in this group, device was used to provide vibration. The device, at room temperature, was placed by the researcher on the peripheral intravenous catheterization application area before the application was performed. For one minute before the application, a slight, non-discomforting vibration was applied to the intervention area.
  Interventions: Other: Vibration Application
- The control group (No Intervention): No intervention was performed on the control group before the peripheral intravenous catheterization procedure, and the standard peripheral intravenous catheterization procedure was performed.

INTERVENTIONS:
Other: Cold Application — Before peripheral intravenous catheterization, heat of approximately 40-42 o C was applied for 1 minute to the area of the procedure using a hot pack, which is one of the dry heat application methods. The heat application pack has a feature that it can maintain its temperature when taken out of hot water and does not disturb the person when it comes into direct contact with the skin. In order to apply heat to the individuals in this group, a pack of 11 x 19 cm is used. This pack is covered with cloth and contains a non-toxic gel, and is placed in hot water to prepare it for use. Because this pack is reusable, it was disinfected before and after each use.
  Arms: Cold Application Group
Other: Heat Application — Before peripheral intravenous catheterization, heat of approximately 40-42 o C was applied for 1 minute to the area of the procedure using a hot pack, which is one of the dry heat application methods. The heat application pack has a feature that it can maintain its temperature when taken out of hot water and does not disturb the person when it comes into direct contact with the skin. In order to apply heat to the individuals in this group, a pack of 11 x 19 cm is used. This pack is covered with cloth and contains a non-toxic gel, and is placed in hot water to prepare it for use. Because this pack is reusable, it was disinfected before and after each use.
  Arms: Heat Application Group
Other: Vibration Application — With individuals in this group, the Buzzy® device was used to provide vibration. The Buzzy® device, at room temperature, was placed by the researcher on the peripheral intravenous catheterization application area before the application was performed. For one minute before the application, a slight, non-discomforting vibration was applied to the intervention area. As the Buzzy® device can be used more than once, it was disinfected after each use and before being used with another individual. In this study, the body of the device was used, and only vibration was applied to the individuals in this group.
  Arms: Vibration Application Group

SUMMARY:
Aim: The aim of the present study was to examine the effect on venous dilation, procedure duration and pain severity of local hot, cold and vibration applications performed on the intervention area before peripheral intravenous catheterization in adults.

Methods: The study included 120 adults who were randomly selected between March and August 2023. One application group (n=30) received local hot application, one group (n=30) received local cold application, and one (n=30) received local vibration using the Buzzy® device. The applications, to the site of the peripheral intravenous catheterization, lasted one minute. The control group (n=30) the received standard peripheral intravenous catheterization application. The groups' venous dilation was assessed on the vein assessment scale and the level of pain felt during catheterization was assessed using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Being in accordance with time and place
* Being aged between 18 and 65 years
* Being able to evaluate the visual analog scale correctly
* Participating voluntarily in the research.

Exclusion Criteria:

* Not participating voluntarily in the research
* Not fitting the inclusion criteria of the research
* Having a vision or hearing problem
* Having a mastectomy
* Having any illness which could affect pain perception, such as sensory-motor disorder, diabetes, peripheral vascular diseases or peripheral neuropathy
* Having an allergy to heat and cold application
* Having phlebitis, scar tissue, dermatitis, an incision or findings of infection at the place where the intervention was to be performed
* Having taken an analgesic (within the previous six hours) or an anesthetic agent before the peripheral intravenous catheterization procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
pain intensity in mm | 6 months
  A 10-cm vertical VAS was used to evaluate the severity of pain felt by the individuals during the procedure. One end indicated lack of pain and the other the most severe pain possible. Pain severity was evaluated in millimeters.
venous dilation in score | 6 months
  Vein Assessment Scale was used in the study to evaluate individuals' veins. There are five assessment steps: (1) veins are neither visible nor palpable, (2) veins are visible but not palpable, (3) veins are barely visible and palpable, (4) veins are visible and palpable, and (5) veins are clearly visible and easily palpable.
procedure duration in sec | 6 months
  In the stages of the peripheral intravenous catheterization intervention of individuals in the application and control groups, a chronometer was started immediately after an automatic tourniquet was attached to the patient's arm. After catheterization was completed successfully and before the evaluation material was applied, the chronometer was stopped, and the procedure duration was recorded in the form of seconds on the data collection form.

SECONDARY OUTCOMES:
weight | 6 months
  weight in kilograms
height | 6 months
  height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yilmaz E, Yilmaz D. The effect of three different nonpharmacological methods on cannulation success during peripheral intravenous catheter placement in the emergency unit: a randomized controlled trial. BMC Anesthesiol. 2024 Oct 9;24(1):362. doi: 10.1186/s12871-024-02723-2. PMID 39385099